CLINICAL TRIAL: NCT01370798
Title: Local Oestrogen Versus Placebo as Preoperative Treatment in Patients With Severe Hypospadias: Effects on Post-operative Complications.
Acronym: HYPOSPADES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2010.608; 2010-023686-22 (EudraCT Number)
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hypospadias
Keywords: Severe hypospadias; local oestrogen; promestriene; Onlay-tube-onlay urethroplasty; post-operative complications; fistula dehiscence
MeSH Terms: conditions — Hypospadias | interventions — promestriene; Hematologic Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- promestriene (Experimental): Children with severe hypospadias treated with promestriene 1%
  Interventions: Drug: promestriene; Procedure: Urethroplasty; Radiation: Wrist X ray; Procedure: Blood test
- Placebo (Placebo Comparator): Control group, children with severe hypospadias treated with Placebo.
  Interventions: Drug: Placebo; Procedure: Urethroplasty; Radiation: Wrist X ray; Procedure: Blood test

INTERVENTIONS:
Drug: promestriene — Promestriene cream 1%, 1g per day during 2 months, cutaneous application
  Arms: promestriene
Drug: Placebo — Placebo of promestriene cream, 1g per day during 2 months, cutaneous application
  Arms: Placebo
Procedure: Urethroplasty — Onlay-tube-onlay urethroplasty performed by a physician expert of this technique (at least 5 years of practical ability)
Radiation: Wrist X ray — Wrist X ray to follow the degree of bone maturation
Procedure: Blood test — Hormonal dosage: Oestradiol, testosterone, FSH-LH and AMH

SUMMARY:
Hypospadias is a congenital abnormality of the penis that is caused by incomplete development of the anterior urethra. This pathology is one of the most common genital anomalies in paediatric urology .The incidence is reported to be 1 out of 250 live male births and is increasing regularly. The hypospadias surgeries present a high risk of post operative complications requiring re-interventions.

A great part of the post operative complications is related to imperfect healing issues. If androgen stimulation seems to be deleterious, at the opposite, oestrogen could impact positively on the skin healing process. This point leads to the hypothesis that local transcutaneous oestrogen stimulation on the ventral and dorsal penile faces decreases the number of skin healing post-operative defects.

The objective of the study is to assess the effect of oestrogen (applied once daily for 2 months prior to surgery) on the post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Severe hypospadias with a division of the corpus spongiosum behind the midshaft of the penis and for which repair requires a urethral substitution by onlay urethroplasty.
* Subjects operated between 9 and 36 months old.
* Subjects operated in one of the departments of paediatric urology involved in the study.
* Surgery performed by a surgeon with at least 5 years of practical experience in the hypospadias surgery.
* Written informed consent obtained from parents or legal guardians prior to the participation to the study
* All hypospadias aetiology (hormonal, karyotype or genetic)

Exclusion Criteria:

* Refusal to participate
* Subjects with glandular hypospadias
* Subjects aged <9 months or > 36months old at time of surgery.
* Subjects who had prior surgery of penis (circumcision or hypospadias surgery)
* Subjects treated with androgens (Human Chorionic Gonadotrophin or delayed testosterone) within 6 months prior to surgery.
* Intolerance to promestriene or its excipients.
* Not affiliated to a healthy or social security cover.
* Known tumoral risk
* Pure or mixed gonadal dysgenesis (45, X0/46,XY)

Ages: 9 Months to 36 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 244 (Actual)
Dates: Start 2011-05-26 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Number of patient with postoperative urethral fistula and dehiscence | 1 year

SECONDARY OUTCOMES:
Re-intervention related to wound healing | 1 year
  Number of re-interventions for fistula or dehiscence not related to stenosis, in the first year post surgery.
post-surgical complications | 1 year
  Total number and type of post-surgical complications
Re-intervention not related to wound healing | 1 year
  Number of re-interventions not related to wound healing
Hormone measurement | 2 months
  Plasmatic concentrations of Oestradiol, Testosterone, LH, FSH at inclusion and at 2 months (at the end of study treatment)
Bone age evaluation | 14 monthes
  Hand and wrist radiography at inclusion and 1 year after surgery.
Clinical tolerance of the treatment | 14 months
  Number and type of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Mouriquand, Prof, Principal Investigator — HOPITAL FEMME MERE ENFANT CHU DE LYON
Locations (4):
- France (4):
  - Service de Chirurgie Pédiatrique Uro-génitale, Hopital femme Mere Enfant, Bron
  - Hôpital Mère-Enfant, Nantes
  - Hôpital Robert Debré, Paris
  - Hôpital NECKER, Paris

REFERENCES:
- [Result] Gorduza D, Plotton I, Remontet L, Gay CL, El Jani M, Cheikhelard A, Blanc T, El Ghoneimi A, Leclair MD, Roy P, Pirot F, Mimouni Y, Gaillard S, Chatelain P, Morel Y, Kassai B, Mouriquand P. Preoperative Topical Estrogen Treatment vs Placebo in 244 Children With Midshaft and Posterior Hypospadias. J Clin Endocrinol Metab. 2020 Jul 1;105(7):dgaa231. doi: 10.1210/clinem/dgaa231. PMID 32386308